CLINICAL TRIAL: NCT01525147
Title: A Block-randomized, Double-blind, Placebo-controlled, Single-dose Escalating, Phase I Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetics of YHB1411-2 in Healthy Male Volunteers
Brief Title: Phase I Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetics of YHB1411-2 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YHB1411-2-101
Record Dates: First submitted 2012-01-26; First posted 2012-02-02 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Rheumatic Arthritis
MeSH Terms: conditions — Rheumatic Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- YHB1411-2: Level 2 (Experimental): The ratio of Test Drug(YHB1411-2) to Placebo is 4 :1.
  Interventions: Biological: YHB1411-2: Level 2; Biological: Placebo
- YHB1411-2: Level 3 (Experimental): The ratio of Test Drug(YHB1411-2) to Placebo is 13 :2.
  Interventions: Biological: YHB1411-2: Level 3; Biological: Placebo
- YHB1411-2: Level 4 (Experimental): The ratio of Test Drug(YHB1411-2) to Placebo is 4 :1.
  Interventions: Biological: YHB1411-2: Level 4; Biological: Placebo
- YHB1411-2: Level 5 (Experimental): The ratio of Test Drug(YHB1411-2) to Placebo is 4 :1.
  Interventions: Biological: YHB1411-2: Level 5; Biological: Placebo
- YHB1411-2: Level 1 (Experimental): All investigational products are YHB1411-2(This level is pilot study).
  Interventions: Biological: YHB1411-2: level 1

INTERVENTIONS:
Biological: YHB1411-2: Level 2 — IV infusion
  Other Names: Undecided
  Arms: YHB1411-2: Level 2
Biological: YHB1411-2: Level 3 — IV infusion
  Other Names: Undecided
  Arms: YHB1411-2: Level 3
Biological: YHB1411-2: Level 4 — IV infusion
  Arms: YHB1411-2: Level 4
Biological: YHB1411-2: Level 5 — IV infusion
  Other Names: Undecided
  Arms: YHB1411-2: Level 5
Biological: Placebo — IV infusion
  Arms: YHB1411-2: Level 2; YHB1411-2: Level 3; YHB1411-2: Level 4; YHB1411-2: Level 5
Biological: YHB1411-2: level 1 — IV infusion
  Other Names: Undecided
  Arms: YHB1411-2: Level 1

SUMMARY:
A block-randomized, double-blind, placebo-controlled, single-dose escalating, phase I clinical trial to evaluate the safety, tolerability and pharmacokinetics of YHB1411-2 in healthy male volunteers

DETAILED DESCRIPTION:
First in human Study

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers of aged between 20 to 45 years old at the time of screening
2. Volunteers weighing over 50 kg with body mass index between 18.0 ~ 28.0 kg/m2
3. Volunteers who has signed a written informed consent voluntarily, prior to any procedure, using a form that is approved by the local Institutional Review Board after detail explanation of the purpose, contents, and characteristic of the drug

Exclusion Criteria:

1. Have history or presence of clinically significant diseases in liver, kidney, gastrointestinal tract, nervous system, respiratory system, endocrine system, blood•tumor, cardiovascular, urinary system, and mental disorder
2. Presence of current tuberculosis or latent tuberculosis or have history of tuberculosis (confirmed by chest X-ray test or tuberculin skin test)
3. Have active infection such as chronic or topical infection
4. Have history of hospitalization or have received antibiotics due to serious infection within 1 month prior to the first administration
5. Have know hypersensitivity to biologicals
6. Have AST(SGOT) or/and ALT(SGPT) > 1.5 times of normal upper limit at the time of screening
7. Shown positive results in any of HBsAg, HCV Ab, HIV Ab tests
8. Have history of drug abuse or shown positive reaction of drug abuse in urine test at the time of screening
9. Received any biological drugs including monoclonal antibody products or protein drugs within the last 6 months prior to the first administration
10. Participated in any other clinical trials within 2 months prior to the first administration of Investigational Product
11. Have donated whole blood within 2 months prior to the first administration of Investigational Product, or donated blood components or received transfusion within 1 month prior to the first administration of Investigational Product
12. Subject who drink continuously (over 21 units/week, 1 unit = 10 g of pure alcohol) or who cannot quit drinking while hospitalized
13. Smoker (Subject can be enrolled if he/she had quit smoking within 3 months before the first administration of Investigational Product (Day 1))
14. Subject who is judged to be ineligible by principal investigator or sub-investigator according to various reasons including their abnormal test results (clinical laboratory test, chest X-ray test, 12-lead ECG)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety Evaluation | Participants will be followed for the duration of hospital stay(an expected average of 1 week) and out-patient visit for 8 weeks → Specified timepoints in the protocol.
  Adverse Events, Physical examination, ECG, Vital sign, Clinical Laboratory Tests results, Chest X-ray

SECONDARY OUTCOMES:
Pharmacokinetic Evaluation | PK sampling : participants will be followed for the duration of hospital stay(an expected average of 1 week) and out-patient visit for 8 weeks → Specified timepoints in the protocol.
Immunogenicity Evaluation | HAHA measurement(blood sampling): pre-dose and out-patient visit for 8 weeks → Specified timepoints in the protocol.
  1. HAHA (Human anti human antibodies) measurement
  2. Neutralizing Antibody measurement: only if antibody formation has verified

CONTACTS AND LOCATIONS:
Overall Officials: Woo-Seung Huh, MD,PhD., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Irwon-dong, Gangnam-gu, South Korea